CLINICAL TRIAL: NCT03551886
Title: Automated Assessment Using Facial Coding
Acronym: R44DA042640
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2R44DA042640-02 (NIH)
Record Dates: First submitted 2018-05-25; First posted 2018-06-11 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental app (Experimental): This is the Advanced Emotion App that we initially developed in phase 1 and are now enhancing in phase 2.
  Interventions: Behavioral: Advanced Emotion App
- Comparison app (Active Comparator): This is the Basic Emotion App, which is an alternative intervention app that controls for time and attention.
  Interventions: Behavioral: Basic Emotion App

INTERVENTIONS:
Behavioral: Advanced Emotion App — The app is designed to help TAY better recognize their emotions using enhanced features
  Arms: Experimental app
Behavioral: Basic Emotion App — The app is designed to help TAY better recognize their emotions using basic features
  Arms: Comparison app

SUMMARY:
Transition-age youth (TAY) from ages 18-26 are vulnerable to substance substance use disorder (SUD). This developmental period, termed "emerging adulthood" includes leaving home, entering college or working for the first time; and for some, aging out of foster care or state custody, which end at age 18. The emerging-adulthood period is prime for experimentation with substances and the development of SUD, and associated problems. A major challenge for TAY is the capacity to regulate their emotions, given the hormone changes and emotional intensity of this stage of life. Indeed, substance use can be a short-term way to regulate emotion. The importance of ER is identified as a core skill that is critical to the successful transition to adulthood. The initial component of ER, accurate identification of emotion, is itself a major challenge. In the phase 1 project a mobile app was developed that uses automated emotion detection to help TAY better recognize their emotions in relation to SUD. We found positive results in our phase 1 study. Phase 2 will see the continuation of the development of the app features. Phase 2 also includes a randomized controlled trial to evaluate the app among TAY with SUD in their natural environment, such as home, and we will conduct pre- and post-evaluation to compare outcomes between the app condition and a control-app condition. The primary outcomes are substance use and emotion regulation. User satisfaction, feedback at the end of phase 2 and app metrics will also be explored. The app can potentially have major public health and clinical impact. It could help improve TAY's ability to become more aware of emotions and understand them in relation to SUD via emotion-focused technoloy. If the product is successful it could be expanded to other populations.

DETAILED DESCRIPTION:
Transition-age youth (TAY) from ages 18-26 are especially vulnerable to substance use, misuse, and substance use disorder (SUD). This developmental period, termed the "age of instability" and "emerging adulthood" includes tasks such as leaving home, entering college; identifying vocational goals; working for the first time; body and sexuality changes; coalescing with a peer group; and for some, aging out of foster care or state custody, which end at age 18. The emerging-adulthood period is prime for experimentation with substances and the development of SUD, and associated problems such as binge drinking, driving under the influence, accidents, fighting and violence, HIV, gang involvement, suicide and self-harm, and vulnerability to date-rape and other sexual assault. A major challenge for TAY is the capacity to regulate their emotions, given the hormone changes and emotional intensity of this stage of life. Indeed, substance use is often described as a short-term way to regulate emotion and there is a long-standing literature documenting the association between emotion regulation (ER) problems and SUD. The importance of ER is also grounded in the developmental literature in which ER is identified as a core skill that is critical to the successful transition to adulthood. The initial component of ER, accurate identification of emotion, is itself a major challenge, especially for people with SUD as they are often not aware of their feelings or confused about them due to the nature of the disorder as well as mental health disorders that often co-occur with SUD. The phase 1 project developed and evaluated a mobile app that uses exciting new technology (automated emotion detection) to help TAY better recognize their emotions in relation to SUD variables. Highly positive results were found in the phase 1 feasibility / pilot study and are now proposing a phase 2 project to continue this work. In phase 2 the app will continue to be developed based on user experience based on end-user feedback and an expert consultant team. Phase 2 also includes a randomized controlled trial to evaluate the app among TAY with SUD. They will have six weeks to use the app in their natural environment, such as home, and will complete pre- and post-evaluation using validated instrumts to compare outcomes between two conditions: the app condition and a control-app condition. The primary outcomes are substance use and emotion regulation. End-user satisfaction with the app will also be obtained as well as app metrics. The app product could have major public health and clinical impact. It could help improve TAY's ability to become more aware of their emotions and understand them in relation to SUD via an exciting emotion-focused technology innovation. If the product is successful it could also be expanded to other populations. The collaborative team includes experts in SUD, TAY, clinical innovations, technology, and app development.

ELIGIBILITY:
Inclusion Criteria: ages 18-26; outpatient; meets criteria for current SUD based on either verification from a professional or via assessment by our team using DSM-5 criteria; has an iPhone; and is not in an environment that restricts substance use (so that our SUD outcomes will be naturalistic).

Exclusion Criteria:

current uncontrolled psychotic or bipolar disorder as the priority for such clients would be to stabilize them on medication; currently suicidal or violent with intent and/or plan; and/or SUD so severe that detoxification is needed, with any of these criteria reported by the TAY and/or a clinical treater. We will not restrict any treatments, self-help or other care of the TAY.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in emotion regulation | baseline and 6 weeks
  Composite of the Toronto Alexithymia Scale and the Difficulties in Emotion Regulation Scale
Change in substance use | baseline and 6 weeks
  Brief Addiction Monitor

SECONDARY OUTCOMES:
Change in psychiatric symptoms | baseline and 6 weeks
  Brief Symptom Inventory
Change in coping | baseline and 6 weeks
  Coping Self-Efficacy Scale
Change in stress | baseline and 6 weeks
  Perceived Stress Scale
Change in distress tolerance | baseline and 6 weeks
  Distress Tolerance Scale
Change in functioning | baseline and 6 weeks
  BASIS-32

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Najavits, Principal Investigator — Treatment Innovations
Locations (1):
- Lisa Najavits, Newton, Massachusetts, United States